CLINICAL TRIAL: NCT06211972
Title: Personality-Targeted Interventions for Addressing Polysubstance Use Among Opioid-Addicted Clients Undergoing Opioid Agonist Therapy: A Feasibility Study
Brief Title: The Feasibility of the OpiVenture Program for Clients Undergoing Opioid Agonist Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Direction 180 | Nova Scotia Mental Health and Addictions (Unknown); Centre for Research, Education, and Clinical Care of At-Risk Populations (RECAP) (Unknown); River Stone Recovery Centre (Unknown); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other); Université de Montréal (Other); University of New Brunswick (Other)
Responsible Party: Principal Investigator, Sherry Stewart, Principal Investigator, Dalhousie University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1029238
Record Dates: First submitted 2023-12-11; First posted 2024-01-18 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Opioid Use Disorder; Polysubstance Addiction; Substance Use
Keywords: Anxiety sensitivity; Hopelessness; Sensation-seeking; Impulsivity; Personality; Psychosocial Interventions; Feasibility; Opioid Agonist Therapy
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Impulsive Behavior

STUDY DESIGN:
Intervention Model Description: A mixed-methods approach nested in a pre-to-post follow-up design
Masking Description: As there is single group on this study, there is no randomization and masking.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): In this study, there is only one study arm, and all eligible participants will be assigned to a treatment group and will participate in three treatment sessions of the OpiVenture program, in addition to the Opioid therapy agonist treatment they are receiving through the recruiting clinic.
  Interventions: Behavioral: OpiVenture

INTERVENTIONS:
Behavioral: OpiVenture — OpiVenture, a targeted psychosocial intervention, complements opioid agonist therapy for opioid use disorder. Adapted from proven interventions like PreVenture, it unfolds over three sessions. Session one covers introductions, an ice-breaker, trait overview, strengths/limitations discussion, goal setting, and homework. Session two reviews homework, explores coping strategies, weighs alternatives, introduces "hot thoughts," reviews trait-specific hot thoughts, and assigns homework. The concluding session involves reviewing homework, identifying personal hot thoughts, challenging them through a cognitive-behavioral exercise, applying insights to goal setting, and concluding with a wrap-up.

SUMMARY:
The opioid crisis continues its devastating impact on Canada, with over 13,900 deaths recorded between 2016 and 2019. Dangerous prescription opioid usage persists, affecting 12.3% of Canadians in 2018. The crisis has escalated, particularly during the COVID-19 pandemic, resulting in increased mortality rates. While opioid agonist therapy (OAT) is a common treatment, it falls short in addressing concurrent polysubstance use, a prevalent issue in OAT clients. Recognizing the limitations of OAT alone, there is a growing recommendation to supplement it with psychosocial interventions.

The PreVenture program, known for its efficacy in reducing substance use, has been adapted for OAT clients, termed "OpiVenture." This study aims to comprehensively assess OpiVenture's feasibility and limited efficacy within an OAT setting. Utilizing a mixed-methods approach, the study design integrates qualitative and quantitative data collection methods to thoroughly evaluate the program's feasibility and preliminary effectiveness. The focus extends beyond immediate outcomes, encompassing the preparation for future randomized controlled trials, including considerations for sample size calculation and recruitment effectiveness. This research addresses the urgent need for more comprehensive interventions to mitigate opioid use disorder (OUD) and associated morbidity, offering a potential solution to improve OAT retention and reduce mortality rates.

DETAILED DESCRIPTION:
The opioid crisis continues to devastate individuals, families, and communities across Canada. In 2016-19, more than 13,900 opioid-related deaths occurred in Canada. Dangerous patterns of prescription opioid use (e.g., using a prescribed opioid without a prescription, outside of its intended purposes, or in excessive quantities) remain a major health threat. Opioids were prescribed to 12.3% of Canadians in 2018. Non-medical use of prescription opioids is markedly higher in Canada/US than elsewhere in the world. Prescription opioids pose an addiction risk of ~5.5% and cost Canadians ~$3.5 billion in healthcare, productivity, and justice costs pre-pandemic. They also pose a threat through the danger of death by overdose. Rates of hospitalization due to opioid poisoning have increased by 27% in the past 5 years, signaling a worsening of the crisis. Opioid-related mortality had been on a steady rise, reaching epidemic proportions pre-pandemic. Overdose rates have increased 5-fold over the past 20 years. Opioid-related deaths have only increased since the COVID-19 pandemic due to the economic downturn and to disruptions to the drug supply chain through border closures. This has resulted in the use of cheaper and more dangerous substances like the powerful synthetic opioids fentanyl and carfentanyl. Pre-pandemic data link fentanyl with 72% of accidental opioid-related deaths in Canada, an 81% increase from the year prior. Street drugs (e.g., heroin, cocaine) are also increasingly being cut with the cheaper fentanyl, leading to a surge in accidental overdoses. Only 0.08% of seized heroin samples tested positive for fentanyl in 2012, whereas 60.1% tested positive in 2017 - an enormous increase in 5 years. Given the progression and escalation of the opioid crisis, opioid use disorder (OUD) is now one of the greatest challenges facing the Canadian health care system, compounded by the COVID-19 pandemic.

Treatment for OUD generally involves pharmacological treatments such as opioid agonist therapy (OAT) including buprenorphine-naloxone and methadone, both of which are efficacious in treating OUD and widely used in Canada. Rooted in a harm-reduction approach, those undergoing OAT are administered a synthetic opioid agonist, under specific controlled dosages. After stabilization, both methadone and buprenorphine/naloxone have shown efficacy for suppressing opioid use, with higher doses being more effective. More recently, alternative OAT treatment modalities including slow-release oral morphine (Kadian) and injectable opioid agonist therapy (iOAT) have been approved for use in opioid addiction medicine within Canada. OAT is effective at reducing opioid use, overdoses, HIV risk, and criminality.

Limitations of OAT: Unfortunately, OAT alone fails to address other problems common in those with OUD. Clients on OAT frequently present with concurrent use of numerous drugs and with high rates of comorbid alcohol, anxiolytic/sedative, stimulant (cocaine/amphetamines), and cannabis use disorders. As a harm reduction treatment, OAT reduces opioid use; but it does not eliminate all opioid use in all OUD clients. OAT clients' polysubstance use includes risky drug combinations, such as opioids (including methadone) plus benzodiazepines (BZs; a class of sedative/anxiolytic), which greatly increases overdose risk, and interferes with optimal treatment outcomes . Experts recommend avoiding concurrent BZ-opioid prescriptions as one of the main ways to combat the opioid crisis . Some individuals in OAT also continue frequently using other drugs such as alcohol, cannabis, and cocaine, including via injection - a particularly risky administration route . Co-use of alcohol and methadone increases overdose risk and negatively impacts cognitive performance and daily functioning. While findings are mixed, recent studies caution that concurrent cannabis use predicts poorer OAT response. Stimulant co-use predicts HIV risk (stimulants are often injected) and poorer OAT retention . Previous research in three studies (60-138 clients per study) at six clinics across Nova Scotia, New Brunswick, & Quebec, highlight the very high rates of polysubstance use in OAT clients . A consistent finding was the very high endorsement of recent polysubstance use, while clients were on OAT: 29% 'topped up' their OAT with another opioid, 27.5% injected drugs, and 54% used BZs despite their well-documented overdose risk with OAT. While OAT has had positive harm reduction effects for OUD, adjunct psychosocial approaches may curb polysubstance use, increase OAT retention, and reduce overdose, providing new solutions to the opioid crisis.

Psychosocial Treatments Supplementing OAT: Psychosocial treatments for substance use disorder (SUD) employ many techniques, including contingency management, relapse prevention, cognitive behavior therapy (CBT), motivational interviewing, and 12-step facilitation. A recent systematic review showed supplementing OAT with psychosocial interventions led to greater treatment attendance, psychological functioning, and adherence to psychiatric medications, and decreased opioid use, alcohol use, and HIV risk. Recent Canadian guidelines for managing OUD released by Canadian Research Initiative on Substance Misuse (CRISM) network, strongly endorse adding psychosocial treatment options to pharmacological interventions, and advocate exploring additional non-pharmacotherapy interventions to supplement OAT. The Opioid Task force of the Canadian Psychological Association recently made similar recommendations and called for increased research in this area to fill important gaps in knowledge around psychosocial and harm reduction interventions that work well in combination with OAT. Despite the availability of psychosocial treatments to supplement OAT, rates of concurrent polysubstance use remain exceedingly high among OAT clients. OAT clinics feel unprepared to deal with complex psychiatric comorbidity and the effective psychosocial interventions require training backgrounds that are not often practical in OAT clinics (e.g., minimum Masters' degree in a mental health field to practice CBT . Interventions that specifically and effectively target concurrent polysubstance use and psychiatric comorbidity are needed to improve OAT retention, particularly those that are developed using a patient-oriented approach to increase their acceptability to patients and are practical for application by OAT service providers to ensure their sustainability in clinics.

Personality Model of Substance Use & Intervention Development: An efficacious and effective protocoled, psychosocial intervention for targeting polysubstance use over the past few decades has been developed, ] and is adaptable to the OAT context providing a possible avenue for additional, acceptable, and sustainable psychosocial treatment that effectively targets clients' dangerous concurrent polysubstance use to improve OAT retention. The personality model of substance use posits that individual differences in substance use patterns are explained by differential sensitivity to the reinforcing effects of alcohol and other drugs, based on functionally distinct motivational systems that are manifested as different traits. Substance use behaviors can therefore be understood through two broad domains of personality - the disinhibited (i.e., externalizing) and inhibited (i.e., internalizing) domains - which in turn can be broken down into four lower-order personality traits that are intimately linked with substance use. Elevations on these four personality traits have been shown to predict risk for using specific substances, differential motivational profiles for substance use , differential sensitivity to the pharmacological effects of various drugs, and vulnerability to co-morbid psychiatric disorders.

Using a combination of motivational enhancement and cognitive-behavioral skills-building via in-session group activities and homework, these interventions target specific personality-relevant cognitive distortions (see below) and have been repeatedly shown to delay or reduce alcohol and other substance use by 30-80% among high-risk youth.

Within the disinhibited domain, lower-order personality traits associated with substance use are sensation seeking (SS; novelty/pleasure seeking) and impulsivity (IMP; disinhibited personality). Within the inhibited domain, lower-order traits associated with substance use are anxiety sensitivity (AS; fear of arousal) and hopelessness (HOP; depression proneness). These traits can be quickly measured with the widely validated, and internationally used Substance Use Risk Profile Scale (SURPS). Within the four-factor model of substance use, sensation seeking is characterized by a preference for novel and exciting activities, and by boredom proneness.

A Framework for Validation, Intervention Adaptation and Testing: Due to the clear need for more effective psychosocial interventions to supplement OAT for addressing OUD and related morbidity, the ongoing high rates of polysubstance use among OAT clients, and extremely high rates of OAT dropout, PreVenture and CoVenture has been adapted to OUD clients in the OAT clinic context, and is being called "OpiVenture". The framework underlying OpiVenture's development is the U.S. National Institute of Health's (NIH's) ORBIT model for psychosocial and behavioral treatment development. This evidence-based framework centers around a stakeholder-informed significant clinical research question: "How can dangerous patterns of polysubstance use be curbed and how can OAT retention improve to reduce morbidity and mortality?" The ORBIT model provides guidance through four phases for improving the systematic development, adaptation, and testing of appropriately designed and innovative psychosocial interventions. In Phase I, the intervention is designed based on evidence from basic behavioral and psychosocial research and stakeholder input. In Phase II, preliminary testing of the intervention takes place (e.g., feasibility studies). It is only after Phases I-II that one proceeds on to Phases III-IV: Efficacy (RCTs) and Effectiveness (trials under real world conditions), returning to earlier phases for refinement as necessary. A patient-oriented integrated knowledge translation (iKT) approach is embedded throughout to ensure that developed interventions are acceptable to patients and practitioners.

Phase I of OpiVenture development has been completed investigating the role of personality in the maintenance of substance use among OAT clients, validating the four-factor personality model in this client demographic. Using qualitative interview data focused on clients' understanding of their personality, substance use patterns, contexts, and triggers for their substance use, has informed the adaptation of existing personality-targeted intervention manuals. Additionally, focus groups with OAT clinic service providers and staff informed intervention delivery format, including ideal contextual parameters such as scenarios and session lengths.

ELIGIBILITY:
Inclusion Criteria:

Currently enrolled in Opioid Agonist Therapy at one of the 4 partner clinics in Quebec and Atlantic Canada for 30 days

≥18 years of age Score at least one standard deviation (SD) above the population-specific norm on 1 of 4 personality traits on the Substance Use Risk Profile Scale (SURPS ) Ability to understand spoken English or French Ability to provide informed consent

Exclusion Criteria:

Those who are unable to provide informed consent and indicate severe cognitive impairment -measured by the Mini-Mental State Examination (MMSE), will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of substance-using days | Baseline, one-month follow up, and four-month follow up
  This outcome will be measured by self-report data collected via timeline-follow back (TLFB) assessment which uses a calendar to examine substance use in detail for each day in the past 30, starting with the most recent event
Retention of participants in the Opioid Agonist Therapy Program | Baseline, one-month follow up, and four-month follow up
  If a client is not available for a 1- or 4-month follow-up assessment, we will check with the clinic's database to determine if this client is still receiving OAT services at the clinic. If they are no longer receiving OAT services, they will be defined as an OAT dropout for the purposes of retention analyses

SECONDARY OUTCOMES:
Changes in mental health of study participants | Baseline, one-month follow up, and four-month follow up
  Using the 21-item Depression, Anxiety and Stress Scale (DASS-21), we will measure changes in depression, anxiety and stress over time. The DASS-21 is the short form of the DASS-42, a self-report scale designed to measure the negative emotional states of depression, anxiety and stress. The minimum and maximum values for each subscale are as follows: depression (0-21), anxiety (0-21), and stress (0-21). Higher scores indicate greater severity of symptoms.
The risky, impulsive, and self-destructive behaviors | Baseline, one-month follow up, and four-month follow up
  To measures risky, impulsive, and self-destructive behaviors, we will use the 38-item The Risky, Impulsive, & Self-destructive behavior Questionnaire (RISQ). The RISQ is a self-report questionnaire that assesses a wide range of behaviors, including substance use, aggression, and self-harm. The scale has a minimum score of 0 and a maximum score of 114, with higher scores indicating more risky, impulsive, and self-destructive behaviors.
Motives for substance use questionnaire | Baseline, one-month follow up, and four-month follow up
  To measure clients' motives for substance, we will use the Substance Use Motives Measure (SUMM). The SUMM is an eight-factor model that identifies eight motives for alcohol and substance use: Enhancement, Social, Conformity, Anxiety-Coping, Depression-Coping, Boredom-Coping, Self expansion, and Performance. Higher scores on the SUMM indicate a greater endorsement of the motives for substance use.
Participants' changes in subjective pain | Baseline, one-month follow up, and four-month follow up
  Subjective pain will be measured by Short Form McGill Pain Questionnaire II (SF-MPQ-II) and enhanced Chronic Pain Questionnaire (eCPQ) . The SF-MPQ-II is a shorter version of the original McGill Pain Questionnaire (MPQ) and assesses the major symptoms of both neuropathic and non-neuropathic pain. It includes 22 items with 0-10 numerical response options. Higher scores on the SF-MPQ-II indicate a greater intensity of pain, while higher scores on the eCPQ indicate a greater impact of chronic pain on an individual's life
Participants' changes in subjective pain | Baseline, one-month follow up, and four-month follow up
  Subjective pain will be measured by the enhanced Chronic Pain Questionnaire (eCPQ) as well . The eCPQ module comprises 14 items that evaluate the presence of chronic pain (defined as pain that persists for ≥3 months, beyond the normal time of healing) and assess pain intensity, location, and pain-related interference with function, sleep, and mood . Higher scores on the eCPQ indicate a greater impact of chronic pain on an individual's life.

OTHER OUTCOMES:
Socio-Demographic Questionnaire. | At baseline
  We will collect sociodemographic data including age, sex, gender identity, ethnicity, socio-economic status, living circumstances, relationship status, education and Opioid Agonist Therapy history including current type of Opioid Agonist Therapy and dose, clinic, pain
Personality Traits | At baseline
  Personality will be assessed with the reliable and valid 23-item Substance Use Risk Profile Scale (SURPS). The SURPS has 4 subscales which each tap one personality factor in the 4-factor model . Comparisons of respondents' scores on these measures relative to norms will be used for selection into OpiVenture and for assignment to a specific intervention (i.e., Anxiety Sensitivity, Hopelessness, impulsivity, or Sensation-seeking).Higher scores on the SURPS subscales indicate a higher likelihood of substance use.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Stewart, PhD, Principal Investigator — Dalhousie University

IPD SHARING:
Plan to Share IPD: No